CLINICAL TRIAL: NCT06072469
Title: Comparison of Shoulder Range of Motion and Isometric Strength Before and After a Single Badminton Match in Young Elite Badminton Players of Rawalpindi.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yusra Medical and Dental College (Other)
Responsible Party: Principal Investigator, Maham Nasir, Head of Physical Therapy Department, Yusra Medical and Dental College
Other Study IDs: ROM
Record Dates: First submitted 2023-09-18; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Athletes
Keywords: ROM; Isometric Strength; Single Match

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to compare the result of shoulder ranges of motion and isometric strength before and after a single badminton match in young elite badminton players of Rawalpindi. This is an observational study. The main questions it aims to answer is; Does the shoulder ranges of motion and isometric strength increases or decreases before and after a single badminton match. ROM and Isometric strength will be performed on the participants.

DETAILED DESCRIPTION:
Badminton is a worldwide popular racquet sport. In badminton, the player uses a variety of multidirectional movement patterns quickly in succession to execute defensive/counterattacking retrievals or construct offensive plays. Although badminton is considered a relatively safe sport, shoulder injuries are very common among both recreational and competitive players.

Badminton injuries are most common of all sports injuries. To meet the functional requirements of their particular activity, overhead athletes need to maintain a careful balance of shoulder mobility and stability. It has been noted that overhead athletes have altered shoulder mobility, which is assumed to arise from adaptive structural alterations to the joint brought on by the high physiological demands of overhead activity.

The scapulothoracic articulation and the glenohumeral joint make up the shoulder complex, which divides the range of motion and increases it. This composition places the glenoid beneath the humeral head to support some of the arm's weight, allowing the implicated muscles to perform in the most productive portion of their length-tension curve.

In the scientific literature, studies on injuries and trauma related to badminton predominate however, some authors report that there are few scientific studies on the relationship between non-serious injuries such as overuse injuries and the history of shoulder pain. Shoulder pain is a very common musculoskeletal complaint in recreational, national, and international competitive players.

Shoulder instability encompasses a spectrum of diseases ranging from subluxation to frank dislocation. While a lot of instability occurrences happen after trauma, instability can also result through recurrent attenuation of the capsuloligamentous structures near the shoulder.

During subluxation, the humeral head translates beyond normal physiological limits, but maintains contact with the glenoid, often resulting in translation to, but not beyond the glenoid rim. While subluxation is often overlooked, it can be problematic, especially in overhead athletes.

Shoulder girdle motion is complex and involves synchronous movement of the scapula, clavicle, and humerus. Two-dimensional (2D and more recently three dimensional (3D) measurement techniques have been used to describe this motion. As the arm is raised, the generally accepted pattern of motion at the shoulder is as follows; the scapula upwardly rotates, posteriorly tilts, and externally rotates; the clavicle elevates and retracts; and the humerus elevates and externally rotates. This coordinated motion, which is reliant on capsulo-ligamentous structures and neuromuscular control, is crucial for the shoulder girdle's correct operation.

There is currently insufficient research on the causes of shoulder pain in badminton players, as far as we could find in our search. Increased age, shorter height, hard training intensity, and more training hours per week, were found to be risk factors for shoulder pain in studies on other overhead motion sports, such as baseball.

There is very limited research purely investigating the short-term effect of overhead play such as single badminton matches. Hence, this study aims to analyze the effects of a single badminton match on young elite players of Rawalpindi and how it affects day-to-day shoulder movement in players.

ELIGIBILITY:
Inclusion Criteria:

* No prior history of shoulder injury or immobility.
* Only elite badminton players
* Players between the age of 16-30 years only.
* Both male and female players.

Exclusion Criteria:

* Participants that have any prior surgical history of the upper limb.
* Participants who play other sports along with badminton.
* Players having any nerve injury or brachial plexus injury.
* Individuals who have systemic joint disease.

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: We are taking the badminton players with no prior history of shoulder injury or immobility, only elite badminton players, players that are between the age of 16-30 years only and both male and female players.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2023-12-28 (Estimated); Study Completion 2024-02-26 (Estimated)

PRIMARY OUTCOMES:
Shoulder Range of Motion | 1 week
  Shoulder range of motion (ROM) refers to the ability of the shoulder joint to move through its full and natural range of movement. A goniometer is one of the widely used instruments for measuring the ranges of motion. The angle obtained by lining up the goniometer's arms with bony landmarks accurately depicts the angle formed by the proximal and distal bones that make up the joint.
  The normal range for shoulder internal rotation is: 0-70 degrees, external rotation: 0-90 degrees , abduction: 0-180 degrees , adduction: 180-0 degrees , flexion:0-180 degrees , extension: 0-60 degrees.
Shoulder Isometric Strength | 1 week
  Manual muscle testing is used for testing the muscle strength. There are total 6 grades of manual muscle testing; 0-5.
  0 indicates no visible contraction, 1 indicates visible palpation without motion, 2 indicates full range of motion with gravity eliminated, 3 indicates full range of motion against gravity, 4 indicates full range of motion against gravity and moderate resistance, 5 indicates full range of motion against gravity with maximal resistance.

CONTACTS AND LOCATIONS:
Locations (1):
- Maham Nasir, Rawalpindi, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fu L, Ren F, Baker JS. Comparison of Joint Loading in Badminton Lunging between Professional and Amateur Badminton Players. Appl Bionics Biomech. 2017;2017:5397656. doi: 10.1155/2017/5397656. Epub 2017 Jun 13. PMID 28694684
- [Background] Chua MT, Chow KM, Lum D, Tay AWH, Goh WX, Ihsan M, Aziz AR. Effectiveness of On-Court Resistive Warm-Ups on Change of Direction Speed and Smash Velocity during a Simulated Badminton Match Play in Well-Trained Players. J Funct Morphol Kinesiol. 2021 Sep 27;6(4):81. doi: 10.3390/jfmk6040081. PMID 34698234
- [Background] Hoskin AK, Watson S, Kamalden TA. Badminton-related eye injuries: a systematic review. Inj Prev. 2023 Apr;29(2):116-120. doi: 10.1136/ip-2022-044564. Epub 2022 Dec 23. PMID 36564168
- [Background] Cejudo A. Risk Factors for, and Prediction of, Shoulder Pain in Young Badminton Players: A Prospective Cohort Study. Int J Environ Res Public Health. 2022 Oct 12;19(20):13095. doi: 10.3390/ijerph192013095. PMID 36293672
- [Background] DeFroda SF, Goyal D, Patel N, Gupta N, Mulcahey MK. Shoulder Instability in the Overhead Athlete. Curr Sports Med Rep. 2018 Sep;17(9):308-314. doi: 10.1249/JSR.0000000000000517. PMID 30204635
- [Background] Fernandez-Fernandez J, Lopez-Valenciano A, Garcia-Tormo JV, Cabello-Manrique D, Garcia-Lopez J. Acute Effects of 2 Consecutive Simulated Badminton Matches on the Shoulder Range of Motion and Isometric Strength of Elite Youth Players. Int J Sports Physiol Perform. 2021 Oct 1;16(10):1447-1453. doi: 10.1123/ijspp.2020-0659. Epub 2021 Mar 10. PMID 33691283
- [Background] Conable KM, Rosner AL. A narrative review of manual muscle testing and implications for muscle testing research. J Chiropr Med. 2011 Sep;10(3):157-65. doi: 10.1016/j.jcm.2011.04.001. Epub 2011 Aug 9. PMID 22014904
- [Background] Couppe C, Thorborg K, Hansen M, Fahlstrom M, Bjordal JM, Nielsen D, Baun M, Storgaard M, Magnusson SP. Shoulder rotational profiles in young healthy elite female and male badminton players. Scand J Med Sci Sports. 2014 Feb;24(1):122-8. doi: 10.1111/j.1600-0838.2012.01480.x. Epub 2012 May 22. PMID 22616686
- [Background] Borsa PA, Laudner KG, Sauers EL. Mobility and stability adaptations in the shoulder of the overhead athlete: a theoretical and evidence-based perspective. Sports Med. 2008;38(1):17-36. doi: 10.2165/00007256-200838010-00003. PMID 18081365
- [Background] Wilk KE, Obma P, Simpson CD, Cain EL, Dugas JR, Andrews JR. Shoulder injuries in the overhead athlete. J Orthop Sports Phys Ther. 2009 Feb;39(2):38-54. doi: 10.2519/jospt.2009.2929. PMID 19194026
- [Background] Kent BE. Functional anatomy of the shoulder complex. A review. Phys Ther. 1971 Aug;51(8):947. No abstract available. PMID 4997967
- [Background] Halder AM, Itoi E, An KN. Anatomy and biomechanics of the shoulder. Orthop Clin North Am. 2000 Apr;31(2):159-76. doi: 10.1016/s0030-5898(05)70138-3. PMID 10736387
- [Background] Abrams GD, Renstrom PA, Safran MR. Epidemiology of musculoskeletal injury in the tennis player. Br J Sports Med. 2012 Jun;46(7):492-8. doi: 10.1136/bjsports-2012-091164. Epub 2012 May 25. PMID 22554841
- [Background] Ebaugh DD, McClure PW, Karduna AR. Effects of shoulder muscle fatigue caused by repetitive overhead activities on scapulothoracic and glenohumeral kinematics. J Electromyogr Kinesiol. 2006 Jun;16(3):224-35. doi: 10.1016/j.jelekin.2005.06.015. Epub 2005 Aug 24. PMID 16125416
- [Background] Tate A, Turner GN, Knab SE, Jorgensen C, Strittmatter A, Michener LA. Risk factors associated with shoulder pain and disability across the lifespan of competitive swimmers. J Athl Train. 2012 Mar-Apr;47(2):149-58. doi: 10.4085/1062-6050-47.2.149. PMID 22488280
- [Background] Fahlstrom M, Soderman K. Decreased shoulder function and pain common in recreational badminton players. Scand J Med Sci Sports. 2007 Jun;17(3):246-51. doi: 10.1111/j.1600-0838.2006.00562.x. Epub 2006 Jun 19. PMID 16787446